CLINICAL TRIAL: NCT01617993
Title: Eeva Continued Access Study.
Brief Title: Eeva™ Continued Access Study: Assessing the Usability of Eeva in a Clinical Setting
Acronym: CAS
Status: Completed | Type: Observational
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-AUX-002
Record Dates: First submitted 2012-06-08; First posted 2012-06-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Infertility
Keywords: in vitro fertilization; assisted reproduction; noninvasive imaging of embryos; time lapse imaging of embryos; traditional morphological grading of embryos; prediction of blastocysts; infertility; Genital Diseases, Male; Genital Diseases, Female
MeSH Terms: conditions — Infertility; Genital Diseases, Male; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women undergoing IVF treatment: Women undergoing IVF treatment

SUMMARY:
User questionnaire of Eeva System usability and reports of device malfunctions.

DETAILED DESCRIPTION:
This study is designed to evaluate the use of Eeva by IVF laboratory staff during routine procedures. The fertilized eggs will be placed in an Eeva dish and the development of the embryos will be monitored by the Eeva system in a standard incubator. On day 3 of embryo culture, Eeva blastocyst prediction data will be printed from the system to be used to assist the embryologist in selecting the best embryo(s). The performance of the system will be summarized and the user feedback from the embryologists will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing fresh in vitro fertilization treatment using their own eggs or donor eggs
* Subject is ≥ 18 and ≤ 40 years of age.
* Subject has basal antral follicle count (AFC) ≥ 8 prior to stimulation cycle.
* Fertilization using only ejaculated sperm (fresh or frozen) - no surgically retrieved sperm.
* Subject has ≥ 5 normally fertilized eggs (2 PN)
* Willing to have all 2PN embryos monitored by Eeva
* Willing to comply with study protocol and procedures and able to speak English.
* Willing to provide written informed consent.

Exclusion Criteria:

* Reinseminated eggs.
* History of cancer.
* Gestational carriers.
* Planned preimplantation genetic diagnosis or preimplantation genetic screening.
* Previously enrolled in this study
* Concurrent participation in another clinical study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women in the United States who undergo IVF treatment and imaging of their embryos with Eeva.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
User questionnaire of Eeva System usability and reports of device malfunctions. | Participants will be followed through ongoing pregnancy, at approximately 10-12 weeks gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: Shehua Shen, ELD, MD, Study Director — Progyny, Inc.
Locations (3):
- United States (3):
  - Pacific Fertility Center, San Francisco, California
  - Fertility Physicians of Northern California, San Jose, California
  - Reproductive Science Center, San Ramon, California

REFERENCES:
- See also: Auxogyn, Inc. website — http://www.auxogyn.com